CLINICAL TRIAL: NCT06647407
Title: A Parallel-group Prevention, Phase II, Partially Blinded, Multi-stage Study to Investigate the Immunogenicity and Safety of Pentavalent Meningococcal ABCYW Vaccine Formulations Compared With Licensed Meningococcal Vaccines When Administered Alone in Healthy Children (2 to 9 Years of Age) or Concomitantly With Routine Pediatric Vaccines in Toddlers (12 to 15 Months of Age) and Infants (2 Months of Age).
Brief Title: Safety and Immunogenicity of an Investigational Pentavalent Meningococcal ABCYW Vaccine Against Meningococcal Disease in Children, Toddlers, and Infants
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAN00013; 2023-510465-10 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Meningococcal Immunization; Healthy Volunteers
MeSH Terms: interventions — 4CMenB vaccine; Acetaminophen; DTaP-IPV-HB-PRP-T vaccine; Vaxelis; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Rotavirus Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Partially blinded (treatment assignment is blinded between the two investigational formulation groups, and open label between the investigation and the comparator group)
  * Laboratory personnel will be blinded to the treatment assignment
  * Participants, Investigators, and Site staff preparing and administering the study intervention will be unblinded between the MenPenta and comparator groups but will be blinded between the 2 MenPenta groups The Sponsor will be partially blinded. At the time of periodic data reviews, additional measures are put in place to maintain the blind of the study participants for the Sponsor staff. The data review will be conducted on the basis of blinded outputs (where data of the 2 MenPenta groups and the control group will be reviewed in aggregate, without any distinction by group). By design, the Sponsor team will have access to partially blinded data for individual participants (eg, for assessment of SAE)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Stage 1: MenPenta vaccine formulation 1 (Experimental): MenPenta vaccine formulation 1, children 2-9 years of age
  Interventions: Biological: Pentavalent Meningococcal ABCYW vaccine
- Stage 1: MenPenta vaccine formulation 2 (Experimental): MenPenta vaccine formulation 2, children 2-9 years of age
  Interventions: Biological: Pentavalent Meningococcal ABCYW vaccine
- Stage 1: vaccine comparator(s) (Active Comparator): Comparator vaccines: Bexsero + MenQuadfi, children 2-9 years of age
  Interventions: Biological: MenACYW conjugate vaccine; Biological: Meningococcal group B vaccine
- Stage 2: MenPenta vaccine formulation 1 (Experimental): MenPenta vaccine formulation 1 + routine vaccines, toddlers 12-15 months of age
  Interventions: Biological: Pentavalent Meningococcal ABCYW vaccine; Drug: Paracetamol; Biological: DTap-HepB-IPV-Hib vaccine; Biological: Pneumococcal 13-valent conjugate vaccine
- Stage 2: MenPenta vaccine formulation 2 (Experimental): MenPenta vaccine formulation 2 + routine vaccines, toddlers 12-15 months of age
  Interventions: Biological: Pentavalent Meningococcal ABCYW vaccine; Drug: Paracetamol; Biological: DTap-HepB-IPV-Hib vaccine; Biological: Pneumococcal 13-valent conjugate vaccine
- Stage 2: vaccine comparator(s) (Active Comparator): Comparator vaccines: Bexsero + MenQuadfi + routine vaccines, toddlers 12-15 months of age
  Interventions: Biological: MenACYW conjugate vaccine; Biological: Meningococcal group B vaccine; Drug: Paracetamol; Biological: DTap-HepB-IPV-Hib vaccine; Biological: Pneumococcal 13-valent conjugate vaccine
- Stage 3: MenPenta vaccine formulation 1 (Experimental): MenPenta vaccine formulation 1 + routine vaccines, infants approximately 2 months of age
  Interventions: Biological: Pentavalent Meningococcal ABCYW vaccine; Drug: Paracetamol; Biological: DTap-HepB-IPV-Hib vaccine; Biological: Rotavirus vaccine; Biological: Pneumococcal 13-valent conjugate vaccine
- Stage 3: MenPenta vaccine formulation 2 (Experimental): MenPenta vaccine formulation 2 + routine vaccines, infants approximately 2 months of age
  Interventions: Biological: Pentavalent Meningococcal ABCYW vaccine; Drug: Paracetamol; Biological: DTap-HepB-IPV-Hib vaccine; Biological: Rotavirus vaccine; Biological: Pneumococcal 13-valent conjugate vaccine
- Stage 3: vaccine comparator(s) (Active Comparator): Comparator vaccines: Bexsero + Nimenrix + routine vaccines, infants approximately 2 months of age
  Interventions: Biological: MenACYW conjugate vaccine; Biological: Meningococcal group B vaccine; Drug: Paracetamol; Biological: DTap-HepB-IPV-Hib vaccine; Biological: Rotavirus vaccine; Biological: Pneumococcal 13-valent conjugate vaccine

INTERVENTIONS:
Biological: Pentavalent Meningococcal ABCYW vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular (IM)
  Other Names: MenPenta
  Arms: Stage 1: MenPenta vaccine formulation 1; Stage 1: MenPenta vaccine formulation 2; Stage 2: MenPenta vaccine formulation 1; Stage 2: MenPenta vaccine formulation 2; Stage 3: MenPenta vaccine formulation 1; Stage 3: MenPenta vaccine formulation 2
Biological: MenACYW conjugate vaccine — Pharmaceutical form: Solution for injection in vial Route of administration: Intramuscular (IM)
  Other Names: MenQuadfi®
  Arms: Stage 1: vaccine comparator(s); Stage 2: vaccine comparator(s)
Biological: MenACYW conjugate vaccine — Pharmaceutical form: Powder and solvent for injectable solution in a pre-filled syringe Route of administration: Intramuscular (IM)
  Other Names: Nimenrix®
  Arms: Stage 3: vaccine comparator(s)
Biological: Meningococcal group B vaccine — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: Intramuscular (IM)
  Other Names: Bexsero®
  Arms: Stage 1: vaccine comparator(s); Stage 2: vaccine comparator(s); Stage 3: vaccine comparator(s)
Drug: Paracetamol — Pharmaceutical form:Suspension-Route of administration:oral
  Arms: Stage 2: MenPenta vaccine formulation 1; Stage 2: MenPenta vaccine formulation 2; Stage 2: vaccine comparator(s); Stage 3: MenPenta vaccine formulation 1; Stage 3: MenPenta vaccine formulation 2; Stage 3: vaccine comparator(s)
Biological: DTap-HepB-IPV-Hib vaccine — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: Intramuscular (IM)
  Other Names: Hexyon®
  Arms: Stage 2: MenPenta vaccine formulation 1; Stage 2: MenPenta vaccine formulation 2; Stage 2: vaccine comparator(s); Stage 3: MenPenta vaccine formulation 1; Stage 3: MenPenta vaccine formulation 2; Stage 3: vaccine comparator(s)
Biological: DTap-HepB-IPV-Hib vaccine — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: Intramuscular (IM)
  Other Names: Vaxelis®
  Arms: Stage 3: MenPenta vaccine formulation 1; Stage 3: MenPenta vaccine formulation 2; Stage 3: vaccine comparator(s)
Biological: DTap-HepB-IPV-Hib vaccine — Pharmaceutical form: Oral solution in tube Route of administration: oral
  Other Names: Infanrix hexa®
  Arms: Stage 3: MenPenta vaccine formulation 1; Stage 3: MenPenta vaccine formulation 2; Stage 3: vaccine comparator(s)
Biological: Rotavirus vaccine — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: Intramuscular (IM)
  Other Names: RotaTeq® Rotarix®
  Arms: Stage 3: MenPenta vaccine formulation 1; Stage 3: MenPenta vaccine formulation 2; Stage 3: vaccine comparator(s)
Biological: Pneumococcal 13-valent conjugate vaccine — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: Intramuscular (IM)
  Other Names: Prevnar 13®
  Arms: Stage 2: MenPenta vaccine formulation 1; Stage 2: MenPenta vaccine formulation 2; Stage 2: vaccine comparator(s); Stage 3: MenPenta vaccine formulation 1; Stage 3: MenPenta vaccine formulation 2; Stage 3: vaccine comparator(s)

SUMMARY:
This study is the first study of Sanofi's Pentavalent Meningococcal ABCYW vaccine clinical development program to be conducted in the pediatric population below 10 years of age. The aim of the study is to assess 2 formulations of the MenPenta vaccine compared to licensed meningococcal vaccines when administered alone in children (Stage 1) or concomitantly with routine pediatric vaccines in toddlers (Stage 2) and infants (Stage 3).

Study details include:

The study duration per participant will be up to 12 months for children in Stage 1 and toddlers in Stage 2 and 16 to-19 months for infants in Stage 3.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 9 years (Stage 1) or 12 to 15 months (Stage 2) or 56 to 89 days (Stage 3) on the day of inclusion
* For infants and toddlers, born at full term of pregnancy (≥37 weeks) and with a birth weight ≥ 2.5 Kg or born after a gestation period of period above 28 (> 28 weeks) through 36 weeks with a birth weight ≥ 1.5 Kg and in both cases medically stable as assessed by the investigator, based on the following definition: "Medically stable" refers to the condition of premature infants who do not require significant medical support or ongoing management for debilitating disease and who have demonstrated a clinical course of sustained recovery by the time they receive the first dose of study intervention
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and judgement of the investigator

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months or since birth for infants; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months or since birth for and infants)
* History of any meningitis infection, confirmed either clinically, serologically, or microbiologically
* At high risk of meningococcal infection during the study
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances
* Individual with active tuberculosis
* History of Guillain-Barré syndrome
* For Stage 3 infants: History of intussusception
* Previous vaccination against meningococcal serogroups A, B, C, W, and/or Y with an investigational or marketed vaccine
* For Stage 3 infants: receipt of the first dose of rotavirus vaccine less than 28 days before the first trial vaccination

NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 56 Days to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants with unsolicited immediate adverse events (AEs) | Within 30 minutes after each vaccination
  Unsolicited systemic AEs that occur within 30 minutes after vaccination
Number of participants with solicited injection site reactions or systemic reactions | Within 7 days after each vaccination
  Pre-defined solicited injection site reactions and systemic reactions that are pre-listed in the diary cards and CRF
Number of participants with unsolicited AEs | Within 30 days after each vaccination
  Unsolicited AEs other than solicited reactions
Number of participants with serious adverse events (SAEs) | Throughout the study, from first visit until 180 days after the last vaccination
  SAEs (including adverse events of special interest [AESIs]) reported throughout the study
hSBA meningococcal serogroups A, C, W, and Y antibody titers pre-dose and 30 days after the second and third dose in infant participants | For Stage 3: Day 1, Day 91, Day 301-361, Day 331-391
  hSBA titers ≥ 1:8 post-vaccination (post-second and third dose)
hSBA meningococcal serogroups A, C, W, and Y vaccine seroresponse pre-dose and 1 month after the second and third dose in infant participants | For Stage 3: Day 1, Day 91, Day 301-361, Day 331-391
  Seroresponse defined as post-vaccination titers ≥ 1:16 for participants with pre-vaccination hSBA titers < 1:4 or or postvaccination titers ≥ 4 times the lower limit of quantification (LLOQ) for participants with a pre-vaccination titer ≤ LLOQ or a post-vaccination titer ≥ 4 times the pre-vaccination titer for participants with a pre-vaccination titer ≥ LLOQ
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroups A, C, W and Y pre-dose and 1 month after the second and third dose in infant participants | For Stage 3: Day 1, Day 91, Day 301-361, Day 331-391
  Geometric mean titers (pre-dose and post-second and third dose)
Percentage of participants with hSBA titers more or equal to lower limit of quantification (LLOQ) against each of serogroups A, C, W, and Y pre-dose and 1 month after the second and third dose in infant participants | For Stage 3: Day 1, Day 91, Day 301-361, Day 331-391
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference MenB strains) ≥ 1:4 pre-dose and 1 month after second dose of vaccination against serogroup B, before and 30 days after third dose in infants | For Stage 3: Day 1, Day 91, Day 301-361, Day 331-391
  hSBA titers ≥ 1:4 for reference MenB strains
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference MenB strains) ≥ 1:8 pre-dose and 1 month after the second dose of vaccination against serogroup B, before and 30 days after third dose in infants | For Stage 3: Day 1, Day 91, Day 301-361, Day 331-391
  hSBA titers ≥ 1:8 for reference MenB strains
hSBA meningococcal serogroup B seroresponse pre-dose and 1 month after the second dose of vaccination against serogroup B, before and 30 days after third dose in infant participants | For Stage 3: Day 1, Day 91, Day 301-361, Day 331-391
  Seroresponse defined as a 4-fold increase in hSBA titers
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroup B (reference MenB strains) pre-dose and 1 month after the second dose of vaccination against serogroup B, before and 30 days after third dose in infant participants | Day 01, Day 91, Day 181 and Day 211 (for Stage 3)
  Geometric mean titers (pre-dose and post-second dose) for the reference MenB strains
Percentage of participants with hSBA titers more or equal to lower limit of quantification (LLOQ) against each and all of serogroup B (ref. MenB strains) predose and 1 month after 2nd dose against serogroup B, before and 30 days after 3rd dose in infants | For Stage 3: Day 1, Day 91, Day 301-361, Day 331-391
Percentage of participants with hSBA titers less than LLOQ against all serogroup B (ref. MenB strains) pre-dose and 1 month after the 2nd dose of vaccination against serogroup B, before and 30 days after 3rd dose in infants | For Stage 3: Day 1, Day 91, Day 301-361, Day 331-391
hSBA meningococcal serogroups A, C, W, and Y antibody titers in children and toddlers | For Stage 1 and 2: Day 1, Day 31, Day 181, Day 211
  hSBA titers ≥ 1:8 for serogroups A, C, W, and Y
hSBA meningococcal serogroups A, C, W, and Y vaccine seroresponse in children and toddlers | For Stage 1 and 2: Day 1, Day 31, Day 181, Day 211
  Seroresponse defined as post-vaccination titers ≥ 1:16 for participants with pre-vaccination hSBA titers < 1:4 or or postvaccination titers ≥ 4 times the lower limit of quantification (LLOQ) for participants with a pre-vaccination titer ≤ LLOQ or a post-vaccination titer ≥ 4 times the pre-vaccination titer for participants with a pre-vaccination titer ≥ LLOQ
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroups A, C, W and Y pre-dose and 1 month after the second dose children and toddlers | For Stage 1 and 2: Day 1, Day 31, Day 181, Day 211
Percentage of participants with hSBA titers more or equal to lower limit of quantification (LLOQ) against each of serogroups A, C, W, and Y children and toddlers | For Stage 1 and 2: Day 1, Day 31, Day 181, Day 211
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference MenB strains) ≥ 1:4 in children and toddlers | For Stage 1 and 2: Day 1, Day 31, Day 181, Day 211
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference MenB strains) ≥ 1:8 in children and toddlers | For Stage 1 and 2: Day 1, Day 31, Day 181, Day 211
hSBA meningococcal serogroup B (reference MenB strains) vaccine seroresponse in children and toddlers | For Stage 1 and 2: Day 1, Day 31, Day 181, Day 211
  Seroresponse defined as a 4-fold increase in hSBA titers
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroup B (reference MenB strains) in children and toddlers | For Stage 1 and 2: Day 1, Day 31, Day 181, Day 211
Percentage of participants with hSBA titers more or equal to lower limit of quantification (LLOQ) against each and all of serogroup B (reference MenB strains) in children and toddlers | For Stage 1 and 2: Day 1, Day 31, Day 181, Day 211
Percentage of participants with hSBA titers less than the lower limit of quantification (LLOQ) against all serogroup B (reference MenB strains) in children and toddlers | For Stage 1 and 2: Day 1, Day 31, Day 181, Day 211

SECONDARY OUTCOMES:
hSBA meningococcal serogroup B (additional MenB strains) vaccine seroresponse in children, toddler and infant participants | Stage 1 and 2: Day 1 and Day 211. Stage 3: Day 1, Day 331-391
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (additional MenB strains) ≥ 1:4 in children, toddler and infant participants | Stage 1 and 2: Day 1 and Day 211. Stage 3: Day 1, Day 331-391
  hSBA titers ≥ 1:4 for additional MenB strains
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (additional MenB strains) ≥ 1:8 in children, toddler and infant participants | Stage 1 and 2: Day 1 and Day 211. Stage 3: Day 1, Day 331-391
  hSBA titers ≥ 1:8 for additional MenB strains
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroup B (additional MenB strains) in children, toddler and infant participants | Stage 1 and 2: Day 1 and Day 211. Stage 3: Day 1, Day 331-391
Percentage of participants with hSBA composite seroresponse titers more or equal to LLOQ each and all additional MenB strains in children, toddler and infant participants | Stage 1 and 2: Day 1 and Day 211. Stage 3: Day 1, Day 331-391
Percentage of participants with hSBA composite seroresponse titers less than LLOQ all additional MenB strains in children, toddler and infant participants | Stage 1 and 2: Day 1 and Day 211. Stage 3: Day 1, Day 331-391

CONTACTS AND LOCATIONS:
Locations (39):
- Brazil (2):
  - Hospital das Clínicas da Universidade Federal de Minas Gerais- Site Number : 0760001, Belo Horizonte, Minas Gerais
  - Private Practice - Dr. Nelson Rosário- Site Number : 0760004, Curitiba, Paraná
- Czechia (5):
  - Investigational Site Number : 2030003, Jindřichův Hradec
  - Investigational Site Number : 2030004, Ostrava
  - Investigational Site Number : 2030007, Pilsen
  - Investigational Site Number : 2030008, Prague
  - Investigational Site Number : 2030009, Prague
- Denmark (2):
  - Investigational Site Number : 2080002, Hvidovre
  - Investigational Site Number : 2080003, Odense
- Finland (7):
  - Investigational Site Number : 2460006, Espoo
  - Investigational Site Number : 2460001, Helsinki
  - Investigational Site Number : 2460008, Helsinki
  - Investigational Site Number : 2460005, Jarvenpaa
  - Investigational Site Number : 2460004, Oulu
  - Investigational Site Number : 2460002, Seinäjoki
  - Investigational Site Number : 2460007, Tampere
- Germany (7):
  - Investigational Site Number : 2760008, Herxheim
  - Investigational Site Number : 2760006, Hürth
  - Investigational Site Number : 2760007, Hürth
  - Investigational Site Number : 2760005, Krefeld
  - Investigational Site Number : 2760009, Mönchengladbach
  - Investigational Site Number : 2760004, Schönau am Königssee
  - Investigational Site Number : 2760003, Wolfsburg
- Honduras (3):
  - Investigational Site Number : 3400001, San Pedro Sula
  - Investigational Site Number : 3400002, Tegucigalpa
  - Investigational Site Number : 3400003, Tegucigalpa
- Poland (6):
  - Investigational Site Number : 6160006, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160005, Trzebnica, Lower Silesian Voivodeship
  - Investigational Site Number : 6160001, Lodz, Lódzkie
  - Investigational Site Number : 6160003, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160002, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160004, Siemianowice Śląskie, Silesian Voivodeship
- Spain (3):
  - Investigational Site Number : 7240007, Seville, Sevilla
  - Investigational Site Number : 7240009, Madrid
  - Investigational Site Number : 7240004, Madrid
- United Kingdom (4):
  - Investigational Site Number : 8260004, Exeter, Devon
  - Investigational Site Number : 8260007, London, England
  - Investigational Site Number : 8260009, London, England
  - Investigational Site Number : 8260010, Southampton, Hampshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAN00013 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26148&tenant=MT_SNY_9011